CLINICAL TRIAL: NCT03251313
Title: Recombinant Humanized PD-1 Monoclonal Antibody (JS001) Combined With Gemcitabine and Cisplatin (GP) as First Line Treatment for Triple Negative Breast Cancer patients-a Phase 1 Clinical Trial
Brief Title: PD-1(Programmed Death-1) Antibody +GP as First Line Treatment for Triple Negative Breast Cancer(TNBC) Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Director of the Department of Medical Oncology, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fudan-P1-201701
Record Dates: First submitted 2017-06-07; First posted 2017-08-16 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- JS001 120mg+GP (Experimental): Level 1: JS001 120mg +GP q3w,*6 cycles, then JS001 120mg q3w for maintenance therapy for up to approximately 2 years.
  Interventions: Combination Product: JS001 120mg+GP
- JS001 240mg+GP (Experimental): Level 2: JS001 240mg +GP q3w,*6 cycles, then JS001 240mg q3w for maintenance therapy for up to approximately 2 years.
  Interventions: Combination Product: JS001 240mg+GP
- JS001 480mg +GP (Experimental): Level 3: JS001 480mg+GP q3w,*6 cycles, then JS001 480mg q3w for maintenance therapy for up to approximately 2 years.
  Interventions: Combination Product: JS001 480mg+GP
- GP followed by JS001 (Experimental): sequential treatment: Patients receive 6 cycles of GP without JS001 and then receive JS001 maintenance therapy for up to approximately 2 years. JS001 will be given at RP2D.
  Interventions: Combination Product: GP followed by JS001

INTERVENTIONS:
Combination Product: JS001 120mg+GP — In this arm, JS001 120mg will be given at d1; Gem 1000mg/m2 d2,9; DDP(cisplatin) 75mg/m2 d2
  Arms: JS001 120mg+GP
Combination Product: JS001 240mg+GP — In this arm, JS001 240mg will be given at d1; Gem 1000mg/m2 d2,9; DDP 75mg/m2 d2
  Arms: JS001 240mg+GP
Combination Product: JS001 480mg+GP — In this arm, JS001 480mg will be given at d1; Gem 1000mg/m2 d2,9; DDP 75mg/m2 d2
  Arms: JS001 480mg +GP
Combination Product: GP followed by JS001 — In this arm,Patients receive 6 cycles of GP without JS001 and then receive JS001 maintenance therapy for up to approximately 2 years. JS001 will be given at RP2D.
  Arms: GP followed by JS001

SUMMARY:
This is a Phase I dose escalation trial to assess dose-limiting toxicity (DLT) and MTD of JS001+GP in advanced/metastatic TNBC patients, and to determine the recommended Phase II dose and the best combination regimen.

DETAILED DESCRIPTION:
There will be 3 stages in this trial. Stage 1 is the dose escalation stage. JS001 will be tested in combination with GP in 3 dose levels.

Level 1: 120mg Level 2: 240mg Level 3: 480mg Patients will receive JS001+GP for 6 cycles and JS001 maintenance therapy for up to approximately 2 years.

JS001 will be given on d1 every 3 weeks with GP and every 2 weeks in maintenance therapy.

The first group of participants will receive the lowest dose level of JS001 at 120mg. Each new group will receive a higher dose of JS001 than the group before it until 480mg.

Stage 2 is the dose expansion stage. Dose expansion will be carried out to expand to 12 patients in the highest dose level at which the patient can tolerate well. This dose will also be recommended as phase 2 dose(RP2D).

Stage 3 is the sequential treatment stage. Patients receive 6 cycles of GP without JS001 and then receive JS001 maintenance therapy for up to approximately 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed relapsed or metastatic triple negative breast cancer
* Subjects must have normal organ and marrow function as defined below:
* White blood cell ≥ 3,000/μL, Absolute neutrophil count ≥ 1,500/μL, Hemoglobin ≥ 9.0 g/dl, Platelet count ≥ 100,000/μL
* Total bilirubin ≤1.25 X institutional upper limit of normal , aspartate aminotransferase(AST) ≤ 2.5 X institutional upper limit of normal, alanine transaminase(ALT) ≤ 2.5 X institutional upper limit of normal (For patients with liver metastasis, Total bilirubin ≤1.5 X institutional upper limit of normal , AST ≤5 X institutional upper limit of normal, ALT ≤5 X institutional upper limit of normal)
* Serum creatinine within normal institutional limits
* thyroid-stimulating hormone ,FT3(free triiodothyronine),FT4(Free thyroid hormone) within 0.9 X institutional lower limit of normal to 1.1 X institutional upper limit of normal (Except for patients who had thyroid ectomy)
* Basically normal EKG and left ventricular ejection fraction(LVEF)>50%
* Life expectancy of 6 months or more
* Performance Status 0-1
* Subjects must have at least one measurable disease per RECIST v1.1
* Weight more than 45 Kilogram
* Subjects must have not received chemotherapy in metastatic setting, subjects relapsed 6 months after the completion of adjuvant therapy are eligible
* Subjects must be willing to supply fresh or archive tumor tissue for research purposes
* Subjects must have stopped receiving any anti-cancer treatment (including chemotherapy, curative radiotherapy, and surgery or targeting therapy) for at least 4 weeks.
* Subjects must have stopped receiving systemic immunosuppressive agents for at least 2 weeks.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Subjects with radiographically stable treated brain metastases are eligible but must not have been on steroid therapy for at least 4 weeks
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Gemcitabine, cisplatin or JS001
* Patients who have adjuvant chemotherapy and relapsed within 6 months.
* Pregnant or breastfeeding women are excluded from this study
* Patients with HIV infection, patients with positive HbsAg or HCV(hepatitis C virus)-RNA
* Patients with chronic autoimmune disease
* Patients with prior therapy with antibodies that modulate T-cell function (e.g., anti-PD-1, anti-PD-L1, anti-CTLA-4(Cytotoxic T-lymphocyte-associated protein 4))
* Patients with evidence of active, non-infectious pneumonia
* Patients with a history of tuberculosis
* Patients active infection requiring intravenous systemic therapy
* Severe cardiovascular disease
* Severe gastrointestinal dysfunction (bleeding, infection, obstruction or ≥ grade 1 diarrhea)
* Patients with severe coagulation dysfunction or bleeding tendency, patients who are receiving thrombolysis or anticoagulation therapy
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, severe hyper blood pressure, severe diabetes or severe thyroid disease that would limit compliance with study requirements
* Patients with known psychiatric disorders that would interfere with cooperation with requirements of the trial
* Patients who have received a vaccine within 4 weeks prior to the first dose of JS001
* Patients with a known additional malignancy that is progressing or requires active treatment (within the last 5 years). Exceptions: basal cell carcinoma of the skin, squamous cell carcinoma of the skin or in situ cancers that has undergone potentially curative therapy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of JS001 when combined with GP | 3 weeks
  If 1/6 patients has grade 3 or higher toxicity then escalation proceeds, if 2/6 has grade 3 or greater toxicity then this is declared MTD.

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 85 days
  Cmax of JS001
Area under the plasma concentration versus time curve (AUC) | 85 days
  AUC of JS001
other pharmacokinetics(PK) characteristics of JS001+GP | 85 days
  half life of JS001
Incidence of Treatment-Emergent Adverse Events | 85 days
  Incidence of Adverse Events that need to be treated immediately
Incidence of Severe Adverse Events | 85 days
  Incidence of Adverse Events that cause hospitalization, inability, death, etc
objective response rate of JS001+GP | 1 year
  objective response rate(%) is the sum of CR(complete remission) rate and PR(partial remission) rate
disease control rate of JS001+GP | 1 year
  disease control rate(%) is the sum of CR rate and PR rate and SD(stable disease) rate for more than 6 weeks
duration of regression of JS001+GP | 1 year
  duration of regression(months) is the time interval from randomization to disease progression
time to regression of JS001+GP | 1 year
  time to regression(months) is the time interval from randomization to disease regressin
progression free survival of JS001+GP | 1 year
  progression free survival(months) is the time interval from randomization to disease progression or death from any reason
overall survival of JS001+GP | 1 year
  overall survival(months) is the time interval between randomization and death from any reason
best combination regimen | 1 year
  Is JS001 combined with GP or GP followed by JS001 better in safety (incidence of grade 3-4 toxicity) and efficacy(Response Rate and PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, MD& PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided